CLINICAL TRIAL: NCT04501172
Title: Impact of Spectacles on Compliance to Mask-wearing Directives in Greece
Brief Title: Impact of Spectacles on Compliance to Mask-wearing Directives
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES8/Th5/25-06-2020
Record Dates: First submitted 2020-07-25; First posted 2020-08-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: face masks; spectacles; contact lenses; compliance in mask-wearing directive
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: People who use social networks, with permanent residence in Greece, aged above 18 years old and adequate literacy of Greek language
  Interventions: Behavioral: Questionnaire completion

INTERVENTIONS:
Behavioral: Questionnaire completion — Participants are contacted through social networks (Facebook) which provide a link to website that contains the questionnaire. Then, they complete the questionnaire which consists of the following 2 parts:
  1. participant's demographic characteristics with questions regarding age, visual acuity - refractive error, spectacles and contact lenses use, and compliance to mask-wearing directives.
  2. 20 items that construct 5 subscales: a) near vision (5 items), b) distance vision (3 items), c) ocular discomfort (3 items), d) driving (2 items), e) limitations (3 items), need for help (2 items), work collaboration (1 item), and emotional impact (1 item).
  The impact of spectacles on the compliance of Greek people to mask-wearing directives will be assessed via this questionnaire.

SUMMARY:
Primary objective of this study is to identify the compliance of Greek people in mask-wearing directive and explore potential associations with refractive errors, spectacles and contact lenses use.

DETAILED DESCRIPTION:
Present study aims to identify whether Greek people have complied with mask-wearing directive and to investigate the correlation of outcomes with visual acuity - refractive errors, spectacles and contact lenses use. For the purposes of this research, a questionnaire of 20 items including the following sub scales have been developed: a) near vision, b) distance vision, c) ocular discomfort, d) driving, e) limitations, need for help, work collaboration, and emotional impact

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Adequate literacy of Greek language
* Permanent residence in Greece

Exclusion Criteria:

* Poor knowledge of Greek language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who use social networks, with permanent residence in Greece, aged above 18 years old and adequate literacy of Greek language
Sampling Method: Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | last 3 months
  1. Gender
  2. Age
  3. Use of spectacles (a. no use, b. for distance, c. for near, d. for distance and near)
  4. Use of contact lenses (a. no use, b. rarely, c. frequently, d. almost always)
  5. Belonging to a vulnerable group (1. No, 2. Yes, 3. I don't know)
  6. Binocular Distance Best Spectacle-Corrected Visual Acuity (if it is known) (1. I don't know, 2. <1/10, 3. 1-3/10, 4. 4-6/10, 5. 7-8/10, 6. 9-10/10)
Compliance to mask-wearing directives | last 3 months
  Compliance to mask-wearing directives
  1. Yes, always
  2. Yes, almost always
  3. Sometimes
  4. No, almost never
  5. No, never
Questionnaire subscale: Near vision | last 3 months
  Difficulty in near vision activities (reading a printed document in the workplace or in daily life, reading a document on computer in the workplace or in daily life, reading a message on mobile phone) when using a face mask
  1. No difficulty
  2. Little difficulty
  3. Some difficulty
  4. Great difficulty
  5. I have stopped this activity because of my vision and the use of face mask
  6. I need to remove my face mask
Questionnaire subscale: Distance vision | last 3 months
  Difficulty in distance vision activities (recognizing people on the opposite sidewalk, reading road and shop signs, crossing roads) when using a face mask
  1. No difficulty
  2. Little difficulty
  3. Some difficulty
  4. Great difficulty
  5. I have stopped this activity because of my vision and the use of face mask
  6. I need to remove my face mask
Questionnaire subscale: Ocular discomfort | last 3 months
  Ocular discomfort (tearing sensation, stinging sensation, general discomfort) when using a face mask
  5-point Likert scale (1 = I absolutely agree / 5 = I absolutely disagree)
Questionnaire subscale: Driving | last 3 months
  Difficulty in driving (during day or night, in known or unknown places) when using a face mask
  1. No difficulty
  2. Little difficulty
  3. Some difficulty
  4. Great difficulty
  5. I have stopped this activity because of my vision and the use of face mask
  6. I need to remove my face mask
Questionnaire subscale: Limitation | last 3 months
  Limitation during physical activity, entertainment, social relationships, professional and learning development when using a face mask
  5-point Likert scale (1 = I absolutely agree / 5 = I absolutely disagree)
Questionnaire subscale: Collaboration | last 3 months
  Difficulty in collaboration with colleagues in the workplace when using a face mask
  1. No difficulty
  2. Little difficulty
  3. Some difficulty
  4. Great difficulty
  5. I have stopped this activity because of my vision and the use of face mask
  6. I need to remove my face mask
Questionnaire subscale: Need for help | last 3 months
  Need for help during shopping (supermarket, grocery store, bakery) or in public services (bank etc) when using a face mask
  5-point Likert scale (1 = I absolutely agree / 5 = I absolutely disagree)
Questionnaire subscale: Emotional impact | last 3 months
  Emotional charge when using a face mask
  5-point Likert scale (1 = I absolutely agree / 5 = I absolutely disagree)

SECONDARY OUTCOMES:
Assessment of the relationship between the compliance to mask-wearing directives and the use of spectacles | immediately after the completion of data collection
  Chi-squared test will be performed to assess if the compliance to mask-wearing directives is related to the use of spectacles
Assessment of the relationship between the compliance to mask-wearing directives and the other demographic characteristics | immediately after the completion of data collection
  Chi-squared test will be performed to assess if the compliance to mask-wearing directives is related to the other demographic characteristics
Assessment of the relationship between the compliance to mask-wearing directives and the questionnaire items | immediately after the completion of data collection
  Chi-squared test will be performed to assess if the compliance to mask-wearing directives is related to the 20 questionnaire items and the corresponding subscales (outcome measures 3-10)
Assessment of the relationship between demographic characteristics and the 20 questionnaire items | immediately after the completion of data collection
  Chi-squared test will be performed to assess if demographic characteristics are related to the 20 items of the questionnaire and to the corresponding subscales (outcome measures 3-10)

CONTACTS AND LOCATIONS:
Overall Officials: Labiris Georgios, MD, PhD, Study Chair — Department of Ophthalmolgy, University Hospital of Alexandroupolis, Greece
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece